CLINICAL TRIAL: NCT01371513
Title: Korean's Practice Patterns for Screening PCA(Prostate Cancer) According to PSA(Prostate-specific Antigen) Level
Brief Title: Korean Practice Patterns for Screening PCA(Prostate Cancer)
Acronym: RESPECT
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 113951
Record Dates: First submitted 2011-05-12; First posted 2011-06-10 (Estimated); Last update posted 2017-05-22 (Actual); Status verified 2017-05

CONDITIONS: Neoplasms, Prostate; Prostate Cancer; Benign Prostatic Hyperplasia
Keywords: Serum prostate specific antigen
MeSH Terms: conditions — Prostatic Neoplasms; Prostatic Hyperplasia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- PSA level: more than 2.5ng/ml
  Interventions: Other: continuous screening

INTERVENTIONS:
Other: continuous screening — practice patterns for screening prostate cancer

SUMMARY:
This is to investigate Korean urologist's practice patterns for screening prostate cancer according to PSA level.

DETAILED DESCRIPTION:
This is to investigate Korean urologist's practice patterns for screening prostate cancer according to PSA level.

ELIGIBILITY:
Inclusion Criteria:

* Male with PSA more than 2.5ng/ml from 1 Jan 2008 to 31 Dec 2008

Exclusion Criteria:

* Age less than 40 at PSA screening
* History of drug use which can affect level of PSA within 6months before PSA screening
* Subject who participate any other clinical trial

Min Age: 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with PSA more than 2.5ng/ml in 2008 from urology department of clinic and general hospital
Sampling Method: Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2010-05; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Number of subjects with prostate biopsy | 1year

SECONDARY OUTCOMES:
Number of subjects with prostate cancer | 1year

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Seoul, South Korea